CLINICAL TRIAL: NCT02583633
Title: Transdermal Nitroglycerin and Nifedipine for Managing Preterm Labor: a Randomized Clinical Trial
Brief Title: Transdermal Nitroglycerin and Nifedipine in Preterm Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Payam Peymani, Head Of Biostatistics Department, Health policy Research Center,Shiraz university of Medical Sciences, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ShirazSUMS
Record Dates: First submitted 2015-10-18; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Managing Preterm Labor
MeSH Terms: interventions — Nifedipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group one have received Transdermal nitroglycerin (Active Comparator): transdermal GTN (Schwarz Pharma AG, Monheim, FRG) were prescribed and placed on the patient forearm. Each patch contained 37.4 mg of glyceryl trinitrate which was released in blood stream (10mg/24hour). After one hour of the first patch application, the uterine contractions were evaluated.
  Interventions: Drug: Transdermal nitroglycerin
- Group two have received nifedipine (Active Comparator): For the nifedipine group, nifedipine 5mg softgel (Daana Pharma Co., Tabriz, Iran) was prescribed. In this group, the order of medicine prescription was as below;
  1. One softgel every 20 min (4 doses)
  2. Two softgel every 6 hr (4 doses)
  3. One softgel every 6 hr (4 doses)
  4. One softgel every 8 hr (3 doses) Likewise, the uterine contractions were checked every one hour and if the contraction didn't subside or there was any change in dilation and effacement, the treatment were stopped and another tocolytic were applied.
  Interventions: Drug: nifedipine

INTERVENTIONS:
Drug: Transdermal nitroglycerin
  Arms: Group one have received Transdermal nitroglycerin
Drug: nifedipine
  Arms: Group two have received nifedipine

SUMMARY:
One of the important complications of pregnancy is preterm labor (PTL) and delivery. There are different tocolytic agents to enhance the time of delivery. The aim of this study was to compare the effect of transdermal nitroglycerin (glyceryl trinitrate, GTN) and oral nifedipine for managing preterm labor. This was a randomized clinical trial in women admitted with diagnosis of PTL. Group one have received transdermal GTN whereas group two have received oral nifedipine, vital signs, FHR, contractions, dilation and effacement as well as gestation age at the time of delivery have been monitored and evaluated in both groups of patient. Our main goal has been delay of delivery to have the most beneficial effect of primary corticosteroid administration for fetus.

ELIGIBILITY:
Inclusion Criteria:

* GA between 24 to 34 weeks
* early-onset signs of delivery (≥4 uterine contractions during 20 minutes, ≥1 centimeters (cm) of dilation and effacement over 80%).

Exclusion Criteria:

* maternal or fetal life-threatening conditions which require emergency termination
* multiple pregnancy
* premature rupture of membrane
* fatal anomaly or intra-uterine fetal death
* cervical dilation ≥4 cm
* any tocolytic treatment in previous days and positive allergy to GTN

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Time of Delivery | Delivery

SECONDARY OUTCOMES:
APGAR scores | Delivery
  The Apgar scale is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. The five criteria are summarized using words chosen to form a backronym (Appearance, Pulse, Grimace, Activity, Respiration).
  The Apgar scale is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. The five criteria are summarized using words chosen to form a backronym (Appearance, Pulse, Grimace, Activity, Respiration).

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046